CLINICAL TRIAL: NCT02904993
Title: Prospective Randomized Study Comparing Regional Anesthetic Blocks and Periarticular Infiltration for the Management of Post-operative Pain After Direct Anterior Total Hip Replacement
Brief Title: Study Comparing Regional Anesthetic Blocks and Periarticular Infiltration for the Management of Post-operative Pain After Direct Anterior Total Hip Arthroplasty
Acronym: DA THA pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John M. Redmond, M.D., Orthopedic Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 16-001154
Record Dates: First submitted 2016-05-16; First posted 2016-09-19 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Degenerative Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- L2 paravertebral block (Other): regional anesthetic nerve blocks using an L2 paravertebral block with ropivacaine
  Interventions: Other: L2 paravertebral block
- periarticular injection group (Active Comparator): periarticular local injection into the periarticular soft tissues at the time of hip replacement using a combination of ropivacaine, epinephrine, ketorolac and morphine sulphate (periarticular injection group).
  Interventions: Other: periarticular injection group

INTERVENTIONS:
Other: L2 paravertebral block — nerve block group will receive preoperatively a L2 paravertebral block with indwelling catheter
  Arms: L2 paravertebral block
Other: periarticular injection group — periarticular injection group will receive the injection cocktail towards the end of the total hip replacement prior to skin closure.
  Arms: periarticular injection group

SUMMARY:
To compare two methods of post-operative pain management in patients undergoing total hip arthroplasty. There is a perception that the periarticular injections may not be as effective in controlling post-operative pain.

Both methods are current standard of care. The investigators want to compare the outcomes of each when patients are randomized to one of the methods compared to the other method of post-operative pain control.

ELIGIBILITY:
Inclusion Criteria:

* Subject scheduled for Direct Anterior unilateral total hip replacement
* Weight ≥ 50 and ≤125 kg
* Intact neurological exam
* Cognitively intact with ability to sign consent

Exclusion Criteria:

* Renal insufficiency with creatinine > 1.5 mg/dl
* Allergic to any of the following : Ropivacaine, Epinephrine, Ketorolac, Morphine sulfate, NSAIDs, Tylenol, Neurontin, Morphine, Oxycodone or Dilaudid.
* Subject taking regular narcotic medications prior to surgery (20mg/day Morphine equivalents for >7days)
* Subject with prior open hip surgery who received regional anesthesia or periarticular injection for post op pain management.
* Subject with contraindication for spinal anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes in pain score | post-operative to 7 days
  Static and dynamic post-operative pain scores, measured on a 1 - 10 visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: John M Redmond, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No